CLINICAL TRIAL: NCT00706186
Title: Phase IV Study Safety & Feasibility of Sodium Oxybate in Mild Alzheimer's Disease Patients.
Brief Title: Safety and Feasibility of Sodium Oxybate in Mild Alzheimer's Disease Patients
Acronym: ALD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn by Investigator, protocol in revision
Sponsor: Clayton Sleep Insititute (Industry)
Collaborators: St. Louis University (Other)
Responsible Party: Eric Powell, PhD, Clayton Sleep Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALD Xyrem
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Mild Alzheimer's Disease
Keywords: Mild Alzheimer's; Disease
MeSH Terms: conditions — Disease | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sodium Oxybate — The patient will maintain a dosage of 4.5 g/day for a duration of 7 days leading to Treatment Visit 1. After successful assessment at Treatment Visit 1, the dosage will be increased to 6 g/day for the duration of the trial. At Treatment Visit 2 (day 21), the dosage will be increased to a dosage of 9 g/day, if tolerated by the patient.

SUMMARY:
Eligible patients will undergo this open label initial safety and feasibility study investigating the use of 6 g/day sodium oxybate in mild AD. A total of 5 visits are included with this trial and total subject participation duration of 7-8 weeks. The screening phase will include an initial screening visit and a screening PSG night. After successful screening, subjects will complete a baseline PSG night and undergo a third PSG night to monitor initial safety and compliance with study drug at a dosage of 4.5 g/day of sodium oxybate. Thus the subject will undergo three consecutive nights of PSG in the sleep center. The patient will maintain a dosage of 4.5 g/day for a duration of 7 days leading to Treatment Visit 1. After successful assessment at Treatment Visit 1, the dosage will be increased to 6 g/day for the duration of the trial. At Treatment Visit 2 (day 21), the dosage will be increased to a dosage of 9 g/day, if tolerated by the patient. The remaining visit will occur at 6 weeks after baseline, with Treatment Visit 3 consisting of two consecutive nights of PSG. Participation will be complete after this visit. Phone follow-up will be made at one week post completion visits to assess any wash-out symptoms. Please refer to Figure for flow of the study design.

DETAILED DESCRIPTION:
Screening Visit (Day -14 to -7): To avoid confusion, all study visits will occur at the Clayton Sleep Institute. A spouse or caregiver is required to attend all visits.

During the screening visit potential patients will provide informed consent, which must signed by both the patient and the caregiver, followed by a medical and sleep history and physical, completion of the Morse Fall Scale, CDR scale, and the Mini-Mental Status exam (MMSE), as well as the drawing of clinical labs, collection of urine drug screen, and completion of 12-lead ECG. Mild AD patients must have a previous clinical diagnosis according to established criteria. Review of concomitant medications, stimulant usage, and vital signs will also be recorded. In order to assess for sleep quality, the Pittsburgh Sleep Quality Index (PSQI) will be administered.

Participants who meet study criteria will be asked to continuously wear a wrist actigraph (Actiwatch Score; Mini Mitter Co., Inc, Sunriver, OR) from the screening visit through the baseline visit. Each subject will be instructed to press an event button at bedtime and upon awakening in the morning. Data collection will be in 60 second epochs. A handwritten sleep and caregiver diary will be maintained for the duration of the study period to document daily bedtime, wake time, stimulant usage as well as provide daily estimates of sleep latency, total sleep time, and sleep quality, as well as dosing compliance, adverse events, and behavior.

Baseline Visit (Day 0-2): The baseline visit will occur 1-2 weeks after the screening visit to allow for a medication washout period if needed. Participants will be asked to arrive at the sleep center at 7:30 PM each of the three nights. During the evening of all three testing nights, concomitant medication and stimulant usage and adverse events will be reviewed, as well as gait stability assessment and vital signs performed. Night one will consist of a screening PSG to assess for potential sleep disorders. Patients who do not meet exclusion criteria for sleep disorders after night one will be excluded from the study. Participants will be allowed to leave in the morning after the screening PSG and return that evening. Night two will again consist of a full PSG, with this night serving as baseline data.

Two hours after the completion of the PSG, patients will complete a battery of tests measuring daytime functioning, memory function, and neurobehavioral testing. Measures include the Epworth Sleepiness Scale (ESS), Fatigue Severity Scale (FSS), Clayton Daytime Functioning Scale (CDFS), PSQI, PVT, the National Adult Reading Test- Revised (NART-R), Rey Auditory Verbal Learning Test (RAVLT), Kendrick Object Learning Task (KOLT), and the Cambridge Cognitive Examination (CAMCOG). Following the battery of measurements, a study physician will complete the Clinician's Interview-Based Impression of Severity (CIBIS) during this visit for the mild AD patients and complete the Caregiver Distress Scale (NPI-CDS). Finally, the Instrumental Activities of Daily Living (IADL) questionnaire will be given and completed.

Night three will once again be an all night PSG to specifically monitor and assess compliance and side effects with the first study drug dosage. A dosage of 4.5 g/day of sodium oxybate will be used for this study night and for the first week of treatment. Prior to the PSG the subject and caregiver will be given instructions for the usage of the study drug with the caregiver to assist in the measuring and dosing of the study drug. Following completion of the PSG, enough study drug for one week will be dispensed. The actigraph and sleep/caregiver diary will be collected, with new diaries given to be completed until the next visit. Phone follow-up will be made 3 days later to assess study drug compliance and any adverse events.

Treatment Visit 1 (Day 7): Approximately one week after completion of the baseline visit, the patient and caregiver will return to the sleep center for a daytime visit to assess study drug compliance, adverse events, and caregiver report via the diary and CDS. The study physician, with caregiver input, will complete the Caregiver Clinical Global Assessment of Change (CCGIC) to assess any change in disease severity from baseline. Concomitant medications and stimulant usage, gait stability, and vital signs will be assessed. The battery of daytime functioning, sleep quality, memory and neurobehavioral, and quality of life measures will be administered. Finally, remaining study drug will be collected and new study drug dispensed with instructions to dose at 6 g/day of sodium oxybate provided to the patient and caregiver. A new sleep/caregiver diary will be provided and an actigraph again dispensed to be worn continuously through Treatment Visit 2. Phone follow-up will be made one week later to assess study drug compliance and any adverse events.

Treatment Visit 2 (Day 21): Approximately three weeks after completion of the baseline visit, the patient and caregiver will return to the sleep center for a daytime visit. All procedures and assessments to be performed will be similar to Treatment Visit 1, with the addition of clinical labs collected and a 12-lead ECG performed. Once again, remaining study drug will be collected and new study drug dispensed with instructions to dose at 9 g/day of sodium oxybate provided to the patient and caregiver, pending tolerability of the patient. If patient is unable to tolerate the increased dosage or in the opinion of the investigator there is question of tolerability, the dosage will remain at 6 g/day. The first phone follow-up will be made 3 days post-visit to assess tolerability if the dosage was increased. Once again if tolerability is in question, the dosage may be titrated back to 6 g/day. A new sleep/caregiver diary will be provided. Phone follow-up will be made each week to assess study drug compliance and any adverse events. Finally, the actigraph will dispensed once more around day 30 (either mailed to the patient or picked up from the sleep center) with instructions for the patient to continuously wear the actigraph through the final visit and to press the event button at bedtime and waketime.

Treatment Visit 3 (Day 42): Approximately six weeks after completion of the baseline visit, the patient and caregiver will return to the sleep center for Treatment Visit 3. The patient and caregiver will arrive to the sleep center at 7:30 PM for both nights of PSG testing performed at this study visit. Night one will serve as an adaptation night and night two for data collection. All procedures and assessments to be performed will be similar to Treatment Visit 2, with the battery of assessments following completion of PSG night two. All study medication, sleep/caregiver diaries, and actigraph will be collected. An end of study physical will be performed in conjunction with the other assessments. Active participation in the study will be concluded with this visit. A final follow-up phone call will be made at one week post final study visit to assess any final adverse events, especially as study drug is withdrawn.

ELIGIBILITY:
Study inclusion:

1. Ages 50 to 65 years
2. Diagnosis of mild AD according to NINCDS-ACDRA criteria and a CDR scale score of 1.0 indicating mild dementia
3. May be on approved AI's, but on a stable dose > 3 months prior to baseline and maintain dosage for duration of the study
4. A reliable caregiver, who must reside with the patient, must be present and available for the duration of the study and must attend all study visits and spend the night in the sleep center for Night 3 for the baseline visit. Overnight stays for all other PSG procedures is optional for the caregiver
5. Complaint of sleep disturbance as measured by a score of >5 on the Pittsburgh Sleep Quality Index (PSQI)
6. Fluent in the English language
7. Able to comprehend and comply with all study related procedures

Exclusion Criteria:

1. Previous history and diagnosis of a sleep disorder (such as sleep apnea, periodic limb movements, primary insomnia, or narcolepsy)
2. On screening polysomnogram (PSG) an apnea/hypopnea index (AHI) > 15/hr using CMS criteria, oxygen desaturation < 80%, or periodic limb movement arousal index > 10/hr.
3. Current unstable major medical or psychiatric disorder (unrelated to dementia)
4. A history of succinic semialdehyde dehydrogenase (SSADH) deficiency
5. History of seizure disorder or major affective disorder
6. History of substance abuse
7. Poor gait and coordination
8. Currently taking CNS depressants, stimulants, or other medications in the opinion of the investigator that may affect sleep architecture (other than approved AI therapy). Consistent with study drug labeling, patients taking sedative/hypnotics and unable to washout of those medications at least 7 half-lives prior to completion of initial screening will be excluded.
9. Typically consume > 600 mg caffeine in a 24 hour period and/or unwilling to refrain from caffeine consumption within 4 hours of bedtime
10. Any patient, in the opinion of the investigator, that would not be appropriate for participation in the study

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)

PRIMARY OUTCOMES:
To evaluate and monitor the safety and tolerability of 6 to 9 g/day sodium oxybate in patients with mild Alzheimer's disease (AD) between the ages of 50 and 65 years. | 65 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Powell, PhD, Study Director — Clayton Sleep Institute
Locations (1):
- Clayton Sleep Institute, St Louis, Missouri, United States

REFERENCES:
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083